CLINICAL TRIAL: NCT00071851
Title: A Phase IB Clinical Trial to Evaluate the Safety and Immunogenicity of a Multiclade HIV-1 DNA Plasmid Vaccine, VRC-HIVDNA009-00-VP, Administered at 2 Different Dosing Schedules, in HIV-1-Uninfected Adult Participants
Brief Title: Safety of and Immune Response to an HIV-1 DNA Vaccine (VRC HIVDNA009-00-VP) in HIV Uninfected Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 052; 10198 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2003-11-03; First posted 2003-11-05 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: VRC-HIVDNA009-00-VP

SUMMARY:
The purpose of this study is to test the safety of and immune response to an HIV-1 vaccine, VRC-HIVDNA009-00-VP, in HIV uninfected participants. Two different doses of the vaccine will be tested.

DETAILED DESCRIPTION:
The worldwide HIV epidemic highlights the importance of developing an affordable, globally successful vaccine for HIV prevention. The VRC-HIVDNA009-00-VP vaccine used in this study was developed to incorporate HIV genes from multiple virus clades, representing the viral subtypes responsible for about 90% of new HIV infections in the world. The purpose of this study is to determine the safety and immunogenicity of VRC-HIVDNA009-00-VP in healthy, HIV uninfected individuals.

Participants will be randomly assigned to one of three groups and will be followed for one year. Study injections will be given by needle-free intramuscular injection at the start of study and at Months 1 and 2. Group 1 will receive 3 injections of the study vaccine; Group 2 will receive 2 injections of the study vaccine (at start and Month 2) and injection of placebo (at Month 1); Group 3 will receive 3 injections of placebo. After a screening visit, study visits will occur at enrollment (initial injection) followed by 5 visits every 14 days for the first 2.5 months, with three additional visits at Months 6, 9, and 12. All participants will undergo physical exams, blood and urine tests to assess measures of health, and blood tests to assess HIV infection and immune response to the injections.

ELIGIBILITY:
Inclusion Criteria

* Understanding of vaccination procedure
* Willing to receive HIV test results and provide informed consent
* Good general health
* HIV negative
* Hepatitis B surface antigen negative
* Anti-hepatitis C virus (HCV) antibody negative, or negative for HCV PCR if the anti-HCV is positive
* Not pregnant and agrees to use acceptable forms of contraception

Exclusion Criteria

* HIV vaccines or placebo in a prior HIV vaccine trial
* Immunosuppressive medications within 168 days prior to study
* Blood products within 120 days prior to study
* Immunoglobulin within 60 days prior to study
* Live attenuated vaccines within 30 days prior to study
* Investigational research agents within 30 days prior to study
* Medically indicated subunit or killed vaccines within 14 days prior to study
* Current anti-tuberculosis prophylaxis or therapy
* Anaphylaxis or other serious adverse reactions to vaccines; a person who had an adverse reaction to pertussis vaccine as a child is not excluded
* Autoimmune disease or immunodeficiency
* Active syphilis infection
* Unstable asthma (e.g., use of oral, orally inhaled, or intravenous corticosteroids, emergent care, urgent care, hospitalization or intubation during the past 2 years)
* Diabetes mellitus; a participant with past gestational diabetes is not excluded
* Thyroid disease, including removal of thyroid and diagnoses requiring medication
* Serious angioedema
* Hypertension
* Diagnosis of bleeding disorder
* Malignancy, except those with a surgical excision and subsequent observation period that in the investigator's estimate has a reasonable assurance of sustained cure and/or is unlikely to recur during the period of the study
* Seizure disorder requiring medication within the last 3 years
* Absence of the spleen
* Mental illness that would interfere with compliance with the protocol
* Pregnant or breastfeeding
* Two or more elevated liver function tests

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180
Dates: Start 2003-12; Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie McElrath, Study Chair — Fred Hutchinson Cancer Research Center / University of Washington; Larry Peiperl, Study Chair — San Francisco Department of Public Health / University of California - San Diego
Locations (14):
- United States (14):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - San Francisco Vaccine and Prevention CRS, San Francisco, California
  - Project Brave HIV Vaccine CRS, Baltimore, Maryland
  - Johns Hopkins Bloomberg School of Public Health,Ctr for Immunization Research,Project SAVE-Baltimore, Baltimore, Maryland
  - Brigham and Women's Hosp. CRS, Boston, Massachusetts
  - Fenway Community Health Clinical Research Site (FCHCRS), Boston, Massachusetts
  - Saint Louis Univ. School of Medicine, HVTU, St Louis, Missouri
  - NY Blood Ctr./Union Square CRS, New York, New York
  - HIV Prevention & Treatment CRS, New York, New York
  - Univ. of Rochester HVTN CRS, Rochester, New York
  - NY Blood Ctr./Bronx CRS, The Bronx, New York
  - Miriam Hospital's HVTU, Providence, Rhode Island
  - Vanderbilt Vaccine CRS, Nashville, Tennessee
  - FHCRC/UW Vaccine CRS, Seattle, Washington

REFERENCES:
- [Background] Mascola JR, Nabel GJ. Vaccines for the prevention of HIV-1 disease. Curr Opin Immunol. 2001 Aug;13(4):489-95. doi: 10.1016/s0952-7915(00)00246-6. PMID 11498307
- [Background] Boyer JD, Cohen AD, Vogt S, Schumann K, Nath B, Ahn L, Lacy K, Bagarazzi ML, Higgins TJ, Baine Y, Ciccarelli RB, Ginsberg RS, MacGregor RR, Weiner DB. Vaccination of seronegative volunteers with a human immunodeficiency virus type 1 env/rev DNA vaccine induces antigen-specific proliferation and lymphocyte production of beta-chemokines. J Infect Dis. 2000 Feb;181(2):476-83. doi: 10.1086/315229. PMID 10669329
- [Background] Moore JP, Parren PW, Burton DR. Genetic subtypes, humoral immunity, and human immunodeficiency virus type 1 vaccine development. J Virol. 2001 Jul;75(13):5721-9. doi: 10.1128/JVI.75.13.5721-5729.2001. No abstract available. PMID 11390574
- [Background] Osmanov S, Pattou C, Walker N, Schwardlander B, Esparza J; WHO-UNAIDS Network for HIV Isolation and Characterization. Estimated global distribution and regional spread of HIV-1 genetic subtypes in the year 2000. J Acquir Immune Defic Syndr. 2002 Feb 1;29(2):184-90. doi: 10.1097/00042560-200202010-00013. PMID 11832690
- [Background] Manam S, Ledwith BJ, Barnum AB, Troilo PJ, Pauley CJ, Harper LB, Griffiths TG 2nd, Niu Z, Denisova L, Follmer TT, Pacchione SJ, Wang Z, Beare CM, Bagdon WJ, Nichols WW. Plasmid DNA vaccines: tissue distribution and effects of DNA sequence, adjuvants and delivery method on integration into host DNA. Intervirology. 2000;43(4-6):273-81. doi: 10.1159/000053994. PMID 11251382
- [Derived] Jin X, Morgan C, Yu X, DeRosa S, Tomaras GD, Montefiori DC, Kublin J, Corey L, Keefer MC; NIAID HIV Vaccine Trials Network. Multiple factors affect immunogenicity of DNA plasmid HIV vaccines in human clinical trials. Vaccine. 2015 May 11;33(20):2347-53. doi: 10.1016/j.vaccine.2015.03.036. Epub 2015 Mar 25. PMID 25820067